CLINICAL TRIAL: NCT04992247
Title: A Phase 2A Randomized, Placebo-Controlled Study of Intravenous Allogeneic Adipose-Derived Mesenchymal Stem Cells to Treat Post COVID-19 "Long Haul" Pulmonary Compromise
Brief Title: Study of Allogeneic Adipose-Derived Mesenchymal Stem Cells to Treat Post COVID-19 "Long Haul" Pulmonary Compromise
Acronym: BR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sorrento Therapeutics filed for chapter 11 bankruptcy.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-PLH-201BR
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Covid19
Keywords: covid19; long haul; post-acute covid
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-MSC (Experimental): Allogeneic culture-expanded adipose-derived mesenchymal stem cells (MSCs)
  Interventions: Biological: COVI-MSC
- Placebo (Placebo Comparator): Excipient
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: COVI-MSC — 2, 4 or 6 MSC vials (approximately 15 million cells/vial) will be intravenously infused on Day 0, Day 2, or Day 4 depending on assignment to treatment group.
  Group A: 2 MSC vials infused on D0 and 2 vials of placebo on D2 and D4
  Group B: 2 MSC vials infused on D0 and D2 and 2 vials of placebo on D4
  Group C: 2 MSC vials infused on D0 and D4 and 2 vials of placebo on D2
  Group D: 2 MSC vials infused on D0, D2 and D4
  Arms: COVI-MSC
Biological: Placebo — 6 vials of placebo will be intravenously infused on Day 0, Day 2, or Day 4.
  Arms: Placebo

SUMMARY:
This is a Phase 2a randomized, placebo-controlled study designed to investigate the efficacy, safety and tolerability of COVI-MSC in treating post COVID-19 "long haul" pulmonary compromise.

DETAILED DESCRIPTION:
This is a Phase 2a randomized, placebo-controlled multicenter study designed to investigate the efficacy, safety and tolerability of COVI-MSC in treating post COVID-19 "long haul" pulmonary compromise.

COVI-MSC will be administered intravenously on Day 0, Day 2, and Day 4.

ELIGIBILITY:
Inclusion Criteria:

* Has had prior laboratory-confirmed SARS-CoV-2 infection as determined by an approved polymerase chain reaction (PCR) or an approved antigen test of any specimen
* Has had a recent (within a week) negative SARS-CoV-2 test (an approved PCR or antigen test)
* Has had at least moderate or severe post-COVID-19 pulmonary symptoms for at least 3 months which have resulted in reduced physical functioning compared to pre-COVID-19 status
* Willing to follow contraception guidelines

Exclusion Criteria:

* Clinically improving pulmonary status over the month prior to screening
* Undergone a previous stem cell infusion unrelated to this trial
* Pregnant or breast feeding or planning for either during the study
* Suspected uncontrolled active bacterial, fungal, viral, or other infection
* Any significant medical condition, laboratory value or other illness that in the investigator's opinion would interfere or prevent safe participation in the study
* History of a splenectomy, lung transplant or lung lobectomy
* Concurrent participation in another clinical trial involving therapeutic interventions (observational study participation is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in 6-Minute Walk Distance (6MWD) at Day 60 | Baseline to Day 60
  Change in 6MWD at Day 60

SECONDARY OUTCOMES:
Change in 6MWD at Day 30 | Baseline to Day 30
  Change in 6MWD at Day 30
Relief of symptoms on Day 30 and Day 60 | Baseline to Day 30 and Day 60
  Relief of symptoms on Day 30 and Day 60 based on a categorical Symptom Relief Scale, where 0 = no benefit and 4 = nearly complete benefit
Change in Pulmonary Function | Baseline to Day 30 and Day 60
  Change in pulmonary function at Days 30 and 60, as measured by the single-breath test
Change in oxygenation | Baseline to Day 30 and Day 60
  Change in oxygenation at Days 30 and 60, as measured by the SpO2/FiO2 ratio
Change in biomarker levels | Baseline to Day 60
  Change in biomarker levels: plasma lipocalcin-2, matrix metalloproteinase-7, hepatocyte growth factor

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.